CLINICAL TRIAL: NCT06672406
Title: Effect of Probiotic Lacobacillus Reuterii on Serum Bilirubin Levels in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Nurwahyuni Rachim, dr. Nurwahyuni Rachim, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UH105201003
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Hyperbilirubinemia, Neonatal
Keywords: hyperbilirubinemia; probiotic; Lactobacillus reuterii
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial aims to assess the effect of probiotic Lactobacillus reuteri on serum bilirubin levels in preterm infants. The study will be conducted at NICUs in Makassar, Indonesia, enrolling infants born at 32 to <37 weeks gestation with birth weights of 1000-2499 grams. Forty infants will be randomized to receive either L. reuteri probiotic (5 drops daily for 7 days) or no probiotic. The primary outcome is serum bilirubin levels measured at baseline and after 7 days. Secondary outcomes include incidence of hyperbilirubinemia requiring phototherapy and changes in bilirubin levels in those receiving phototherapy. Blood samples will be collected to measure total and direct bilirubin. This trial will provide evidence on whether L. reuteri supplementation can reduce hyperbilirubinemia severity in preterm infants, potentially informing clinical practice regarding probiotic use as an adjunctive therapy for neonatal jaundice in this vulnerable population.
Who Masked: Participant
Masking Description: The preterm infant subjects and their parents were blinded to whether they received the probiotic intervention or were in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Preterm infants who receive 5 drops of probiotic Lactobacillus reuteri for 7 days
  Interventions: Dietary Supplement: Lactobacillus reuterii
- Control Group (No Intervention): Preterm infants who receive standard care without probiotics

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuterii — Participants in the intervention group received probiotic Lactobacillus reuterii if they received enteral feeding > 30 cc/kgBW. 5 drops of probiotics were given for 7 days in the breast milk or formula milk that did not contain probiotics
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to learn about the effect of probiotic Lactobacillus reuterii on the level of serum bilirubin in moderately and late preterm infants with birth weights 1000 grams to 2499 grams who were admitted to the NICU at Dr. Wahidin Sudirohusodo Hospital, Hasanuddin University Hospital and Cahaya Medika Hospital. The main questions it aims to answer are:

* Are bilirubin levels in preterm infants who received probiotics were lower than those who did not receive probiotics?
* Is the incidence of hyperbilirubinemia requiring phototherapy in preterm infants who received probiotics less than those who did not receive probiotics?

DETAILED DESCRIPTION:
This study aims to investigate the effect of probiotic Lactobacillus reuteri administration on serum bilirubin levels in preterm infants. It is a randomized controlled trial conducted at the Neonatal Intensive Care Units of Dr. Wahidin Sudirohusodo Hospital, Hasanuddin University Hospital and Cahaya Medika Hospital in Makassar, South Sulawesi, Indonesia. The study population includes infants born at 32 to <37 weeks gestational age with birth weights between 1000-2499 grams who are admitted to the NICU. Eligible infants are randomized into two groups - an intervention group receiving probiotic L. reuteri (5 drops daily for 7 days) and a control group not receiving probiotics. The primary outcome is serum bilirubin levels, measured at baseline and after 7 days of intervention. Secondary outcomes include incidence of hyperbilirubinemia requiring phototherapy and changes in bilirubin levels in those receiving phototherapy. Blood samples are collected to measure total and direct bilirubin levels. The study aims to enroll 40 infants (20 per group) to detect a clinically meaningful difference in bilirubin levels between groups. This trial will provide evidence on whether probiotic supplementation with L. reuteri can reduce the severity of hyperbilirubinemia in preterm infants. The results may inform clinical practice regarding the use of probiotics as an adjunctive therapy for neonatal jaundice in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Premature Infants (32 - < 37 weeks gestation)
* Birth weight 1000 - 2499 grams
* Sick infants who are treated in the NICU
* Preterm infants who received enteral feeding > 30 cc/kgBB less than 72 hours after birth, without jaundice or jaundice Kremer 1,2, and 3
* Parents have signed their child's consent to participate in the study

Exclusion Criteria:

* Infants with multiple congenital abnormalities
* Infants with jaundice before 24 hours or having jaundice cremer > 4 less than 72 hours from birth
* Infants with Sepsis, Metabolic acidosis

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Total bilirubin level | Total bilirubin level was measured after 7th day of intervention
  We compare the total bilirubin level between participants who received probiotics and those who did not receive probiotics

OTHER OUTCOMES:
Phototherapy | The need for phototherapy was assessed throughout the intervention (7 days)
  We compare the number of participants who needed phototherapy between probiotic and non-probiotic group

CONTACTS AND LOCATIONS:
Overall Officials: Nurwahyuni Rachim, MD, Principal Investigator — Hasanuddin University
Locations (1):
- Hasanuddin University, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aagaard K, Ma J, Antony KM, Ganu R, Petrosino J, Versalovic J. The placenta harbors a unique microbiome. Sci Transl Med. 2014 May 21;6(237):237ra65. doi: 10.1126/scitranslmed.3008599. PMID 24848255

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT06672406/Prot_SAP_000.pdf